CLINICAL TRIAL: NCT06166966
Title: The Effect of the Flipped Learning on Nursing Students' Asepsis Knowledge and Learning Skills: A Randomized Controlled Study
Brief Title: Use of the Flipped Classroom Model With Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Aysun Acun
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2023-12

CONDITIONS: Use of the Flipped Classroom Model With Nursing Students
Keywords: Flipped training; nursing students; teaching

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- flipped training (Experimental): flipped training
  Interventions: Other: Flipped Education Model
- Course success (Experimental): Course success
  Interventions: Other: Flipped Education Model

INTERVENTIONS:
Other: Flipped Education Model — The effect of the Inside Out Education Model on the course success of nursing students.

SUMMARY:
This study aimed to evaluate the effect of the flipped learning model on the concept of asepsis and learning skills of nursing students. It is aimed to continue teaching the knowledge and skills regarding the subject of flipped teaching outside the classroom. Other goals include raising awareness by focusing on the student, transferring relevant learning to behavior, and students' repeated lessons with videos according to their own learning speed. In the research, students in the experimental group will be shown the principles of asepsis through videos 15 days before the normal course period, and the training will last for four weeks in total. A knowledge test will be administered before and after the training.

DETAILED DESCRIPTION:
The flipped learning model offers students and faculty members the opportunity to teach a course other than the traditional one. It is a blended teaching method in which the activities carried out in the classroom are integrated outside the classroom and the teaching activities carried out outside the classroom are integrated into the classroom. In this model, students can access videos, presentations or recordings prepared as course materials before coming to class, through technological devices such as computers, tablets and smartphones. Students have the opportunity to watch and listen to the prepared course content wherever and whenever they want, as many times as they want. Watching as many resources as they want according to their own learning speed brings about effective and easy learning. Afterwards, when the student comes to the classroom, the information learned is reinforced by the instructor, and the areas that are not understood are solved with questions and answers. Lesson hours for students who take an active role in the classroom are also important in terms of using time effectively. The student is at the center of this learning method and the student assumes individual learning responsibility. Considering nursing education within the scope of all these beneficial results, it is obvious that effective learning will be achieved. This study aimed to help students easily adapt to the principles of asepsis.

Videos containing the principles of asepsis will be presented to the experimental group students 2 weeks before the infection control course (11/11/2023). Normal lecture and practice periods will begin between (11/11/2023-12/12/2023) and the education will last 4 weeks in total. When the study period ends, students will be given a knowledge test and then again 2 weeks later. The implementation period of the study will last until 20/12/2023.

Control group students will be educated only during the normal course. The research will be conducted with first-year students of Bilecik Şeyh Edebali University Nursing Department.

ELIGIBILITY:
Inclusion Criteria: Being a first-year nursing student and receiving training on the concept of asepsis for the first time.

Volunteering to participate in research.

Exclusion Criteria: Students who did not volunteer to participate in the research

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2023-11-11 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
The effect of the Inside Out Education Model on the course success of nursing students. | 11/11/2023-20/12/2023

CONTACTS AND LOCATIONS:
Locations (1):
- Bilecik Şeyh Edebali University, Bilecik, Turkey (Türkiye)